CLINICAL TRIAL: NCT07407608
Title: Single-Dose Image-Guided Radiotherapy (IGRT) With Focal Boost to the MRI-defined Macroscopic Tumor Volume for Intermediate Unfavorable and High Risk Prostate Cancer
Brief Title: ABlative Radiotherapy (for) Unfavorable Prostate Tumors 2.0
Acronym: ABRUPT 2
Status: Recruiting | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Principal Investigator, Stefano Arcangeli, Associate Professor, University of Milano Bicocca
Other Study IDs: ABRUPT 2.0
Record Dates: First submitted 2026-01-29; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer; Prostate Cancer (Adenocarcinoma); Prostate Cancer Non-Metastatic
Keywords: Unfavorable Prostate Tumors; Stereotactic Body Radiotherapy (SBRT); Volumetric Modulated Arc Therapy (VMAT); Prostate Imaging Reporting and Data System (PI-RADS); Toxicity; Quality of Life
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 5 Fx SBRT: Patients will receive 36.25 Gy SBRT in five fractions over two weeks
  Interventions: Radiation: SBRT
- 1 Fx SDRT: Patients will receive 24 Gy SDRT with urethra-sparing and a focal isotoxic GTV boost up to 27 Gy
  Interventions: Radiation: SDRT

INTERVENTIONS:
Radiation: SBRT — Stereotactic Body Radiotherapy. Ultrahypofractionated radiotherapy.
  Groups: 5 Fx SBRT
Radiation: SDRT — Single Dose Radiation Therapy. Ultrahypofractionated radiotherapy.
  Groups: 1 Fx SDRT

SUMMARY:
Published clinical evidence confirms that a single dose of 24 Gy provides unprecedented long-term local control in primary and metastatic prostate cancer with safe toxicity profiles, provided that exposure of surrounding healthy tissues is critically assessed with fulfillment of strict constraints and dose distribution is accomplished using image guidance and tracking tools. In the present trial, intermediate unfavorable and selected high-risk organ-confined prostate cancer patients will undergo Single Dose Radiation Therapy (SDRT) With Focal Boost to the MRI-defined Macroscopic Tumor Volume by means of image-guided volumetric intensity-modulated arc radiotherapy (IGRT-VMAT) and state-of-the-art treatment-planning and quality assurance procedures. Androgen Deprivation Therapy (ADT) type and duration has been set as per standard of care, in accordance with current recommendations and guidelines. The results of the study will enable us to find out if the new, shorter treatment (1 doses of radiotherapy), has a similar level of side effects as the 5 dose treatment and is suitable for further study.

DETAILED DESCRIPTION:
ABRUPT 2.0 is a non-comparative, randomized phase II trial focusing on acute genitourinary (GU) toxicity as the primary endpoint in a similar patient population. Acute GU toxicity was selected because it has been shown to be predictive of late GU toxicity and represents a clinically meaningful early safety endpoint. Using PACE-C as a benchmark, the trial is designed to test the hypothesis that acute GU toxicity in each treatment arm will remain within predefined clinically acceptable limits. Patients are randomized in a 1:1 ratio to receive either 36.25 Gy SBRT in five fractions over two weeks or 24 Gy SDRT with urethra-sparing and a focal isotoxic GTV boost up to 27 Gy. Randomization is performed using a minimization algorithm balanced for NCCN risk group (intermediate-unfavorable vs selected high-risk) and incorporating a random element. Treatment allocation is not masked. All participants are treated at a single institution (Fondazione IRCCS San Gerardo dei Tintori and University of Milan-Bicocca).

All patients undergo non-contrast-enhanced CT and mpMRI simulation on the same day. Anatomic reproducibility is ensured through rectal micro-enema administration. In the SDRT arm, the bladder is filled with 150 mL of saline solution via a 16-F Foley catheter before simulation and treatment delivery. In the five-fraction SBRT arm, bladder preparation consists of drinking 500 mL of still water 30-45 minutes before simulation and each fraction. The use of a hyaluronic acid rectal spacer is encouraged and left at physician's discretion. Patients are positioned supine with arms placed over the chest. CT images and T2-weighted 3D MRI scans are fused for target and OAR delineation. The GTV was defined as the visible tumor lesion on mpMRI in collaboration with an experienced radiologist. The clinical target volume (CTV) encompasses the entire prostate gland and seminal vesicles. The PTV is generated by applying a 3-mm isotropic margin to the CTV. OARs include the urethra, bladder, bladder trigone, rectum, femoral heads, penile bulb, bowel, and neurovascular bundles. In the SDRT arm, a 3-mm isotropic margin is added to the urethra, bladder, and rectum to generate planning OAR volumes (PRV), and the minimum prescribed dose to the GTV and PTV is constrained by OAR dose limits. In the five-fraction SBRT arm, the treatment prescription consists of 36.25 Gy administered in five fractions over two weeks on alternate days, with a mandatory additional CTV dose target of 40 Gy. Both dose levels are prescribed to the isodose covering 95% of the target volume, with controlled dose heterogeneity within the target and a maximum PTV dose of 42 Gy to protect the urethra by limiting its estimated dose to ≤95Gy EQD2. No focal boost is delivered to the GTV in this arm. In both arms, treatment plans are optimized using a 10-MV flattening-filter-free single partial arc (140°-220°), allowing a substantial reduction in treatment time.

In order to preserve identical 3-mm PTV margins in both treatment arms, continuous intrafraction motion monitoring is systematically implemented. Two distinct non-ionizing real-time tracking systems are employed. In the SDRT arm, prostate motion is monitored using an electromagnetic transmitter embedded within a urethral catheter. In the five-fraction SBRT arm, real-time tracking is performed using a 4D transperineal ultrasound system. All treatments are delivered on a linear accelerator. Initial patient positioning is verified using cone-beam CT with soft-tissue matching. Beam delivery is interrupted and patient positioning corrected whenever prostate displacement exceeds 2.5 mm in any of the three spatial directions.

The sample size has been determined using a Simon two-stage minimax design, independently powered for each treatment group to test whether the incidence of acute G2+ toxicity is significantly different from 51% (null hypothesis), using a one-sided 0.05-level test with 90% power to detect a true toxicity rate of 25%. Each group includes 29 patients (stage 1: 25 patients, and stage 2: 4 patients). The trial continued to complete stage 2 as 9 or fewer patients among the first 25 will develop G2+ GU toxicity within 3 months after treatment. If 10 patients or fewer in a group will develop G2+ GU toxicity, this would allow rejecting the null hypothesis of a 51% toxicity rate, which is 1.5 times higher than the rate observed in the PACE-C trial. Under the two-stage design, interim analysis will be provided after 10 patients are treated in each group to ensure that acute toxicity rates are within acceptable limits before proceeding to full accrual. The trial is not powered to detect statistical differences between the two treatment groups; therefore, data will be analysed descriptively.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven prostate adenocarcinoma;
* Intermediate and High risk disease, as per the NCCN definition;
* a PI-RADS 3-5 dominant intraprostatic lesion on multiparametric MRI (mpMRI);
* N0M0 at staging with standard techniques (Bone Scan and Abdominal CT) or (preferably) PSMA PET-CT;
* World Health Organization performance status 0-1;
* Life expectancy of > 5 years, in the opinion of the investigator;
* IPSS score must be ≤ 15 (alpha blockers allowed);
* Prostate gland volume ≤100 g as estimated by computed tomography (CT), ultrasound, or MRI.

Exclusion Criteria:

* ≥T3b disease according to the 8th AJCC classification;
* PSA>20 ng/ml;
* Previous local treatment of the prostate with surgery (radical prostatectomy or cryotherapy) or transurethral resection;
* Previous radiotherapy to the pelvis;
* Presence of a periurethral dominant lesion;
* Previous invasive malignancy unless disease free for a minimum of 5 years;
* Active Crohn's Disease or Ulcerative Colitis;
* Presence of hip prostheses.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unfavorable Intermediate and Selected High Risk Prostate Cancer (no cT3b and PSA > 20 ng/mL allowed), as per NCCN definition
Sampling Method: Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2026-01-28 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2034-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with acute genitourinary treatment-related adverse events as assessed by CTCAE v.5.0 | 3 months
  The primary endpoint is the cumulative incidence of acute CTCAE v5.0 grade ≥2 genitourinary (GU) toxicity from the start of radiotherapy to 3 months post-treatment. Toxicity assessments are performed at baseline, end of treatment, and at 1, 2, and 3 months after radiotherapy.

SECONDARY OUTCOMES:
Number of participants with late genitourinary treatment-related adverse events as assessed by CTCAE v.5.0 | 1, 2 and 5 years
  To assess treatment related late genitourinary (GU) toxicity
Number of participants with treatment-related adverse gastrointestinal events as assessed by CTCAE v.5.0 | 3 months, 1, 2 and 5 years
  To assess treatment related gastrointestinal (GI) acute and late toxicity
QUALITY OF LIFE (QOL) assessed by EORTC QLQ-C30. For QoL domain minimum score (=0) means worst QoL and maximum score (=100) means best QoL. | 3 months, 1, 2 and 5 years
  To measure symptom scores for each QOL domain (overall QoL) by EORTC Questionnaire
Number of participants with voiding symptoms assessed by International Prostatic Symptoms Score (IPSS), ranging from 0 (best) to 35 (worst) | 3 months, 1, 2 and 5 years
  To assess voiding symptoms using IPSS
Number of participants with erectile dysfunction assessed by International Index of Erectile Function Questionnaire ranging from 5 (worst ) to 25 (best) | 2 and 5 years
  To assess erectile function using IIEF 5
Number of participants with biochemical relapse assessed by PSA (Phoenix definition) | 2 and 5 years
  To assess biochemical outcome using serum PSA levels
QUALITY OF LIFE (QOL) assessed by EORTC PR-25. For QoL domain minimum score (=0) means best QoL symptoms and maximum score (=100) means worst QoL symptoms | 3 months, 1, 2 and 5 years
  To measure symptom scores for each QOL domain (urinary incontinence and bowel dysfunction) by EORTC Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Radiation Oncology, Fondazione IRCCS San Gerardo dei Tintori, Monza, MB, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Panizza D, Faccenda V, Ingraito C, Chissotti C, Ferrario F, Colciago RR, De Ponti E, Arcangeli S. Real-time monitoring and appropriate margin selection in linac-based prostate SBRT: Analysis of two different intrafraction motion monitoring systems. Med Phys. 2025 Aug;52(8):e18060. doi: 10.1002/mp.18060. PMID 40802285
- [Background] Panizza D, Faccenda V, Lucchini R, Daniotti MC, Trivellato S, Caricato P, Pisoni V, De Ponti E, Arcangeli S. Intrafraction Prostate Motion Management During Dose-Escalated Linac-Based Stereotactic Body Radiation Therapy. Front Oncol. 2022 Apr 7;12:883725. doi: 10.3389/fonc.2022.883725. eCollection 2022. PMID 35463373
- [Background] Panizza D, Faccenda V, Arcangeli S, De Ponti E. Treatment Optimization in Linac-Based SBRT for Localized Prostate Cancer: A Single-Arc versus Dual-Arc Plan Comparison. Cancers (Basel). 2023 Dec 19;16(1):13. doi: 10.3390/cancers16010013. PMID 38201441
- [Background] Faccenda V, Panizza D, Daniotti MC, Pellegrini R, Trivellato S, Caricato P, Lucchini R, De Ponti E, Arcangeli S. Dosimetric Impact of Intrafraction Prostate Motion and Interfraction Anatomical Changes in Dose-Escalated Linac-Based SBRT. Cancers (Basel). 2023 Feb 10;15(4):1153. doi: 10.3390/cancers15041153. PMID 36831496
- [Background] Draulans C, Haustermans K, Pos FJ, van der Heide UA, De Cock L, van der Voort van Zyp J, De Boer H, Smeenk RJ, Kunze-Busch M, Monninkhof EM, De Roover R, Isebaert S, Kerkmeijer LGW. Stereotactic body radiotherapy with a focal boost to the intraprostatic tumor for intermediate and high risk prostate cancer: 5-year efficacy and toxicity in the hypo-FLAME trial. Radiother Oncol. 2024 Dec;201:110568. doi: 10.1016/j.radonc.2024.110568. Epub 2024 Oct 2. PMID 39362607
- [Background] Tree AC, Hinder V, Chan A, Tolan S, Ostler P, van der Voet H, Kancherla K, Loblaw A, Naismith O, Jain S, Martin A, Price D, Brand D, Chu W, Duffton A, Kelly P, O'Neill B, Staffurth J, Sasso G, Pugh J, Manning G, Brown S, Burnett S, Griffin C, Hall E, van As N; PACE Investigators. Intensity-modulated moderately hypofractionated radiotherapy versus stereotactic body radiotherapy for prostate cancer (PACE-C): early toxicity results from a randomised, open-label, phase 3, non-inferiority trial. Lancet Oncol. 2025 Jul;26(7):936-947. doi: 10.1016/S1470-2045(25)00205-0. Epub 2025 Jun 12. PMID 40517778
- [Background] Arcangeli S, Chissotti C, Ferrario F, Lucchini R, Belmonte M, Purrello G, Colciago RR, De Ponti E, Faccenda V, Panizza D. Ablative Radiation Therapy for Unfavorable Prostate Tumors (ABRUPT): Preliminary Analysis of Toxicity and Quality of Life from a Prospective Study. Int J Radiat Oncol Biol Phys. 2024 Dec 1;120(5):1394-1403. doi: 10.1016/j.ijrobp.2024.06.030. Epub 2024 Jul 4. PMID 38971384